CLINICAL TRIAL: NCT05189054
Title: Safety and Efficacy of SBRT in the Reirradiation for Ultra-central Thoracic Malignant Tumors
Status: Recruiting | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: BYSY-2021-SBRT-UC
Record Dates: First submitted 2021-12-26; First posted 2022-01-12 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-10

CONDITIONS: Stereotactic Body Radiation Therapy; Irradiation; Reaction; Thoracic Tumor; Recurrent Cancer
MeSH Terms: conditions — Thoracic Neoplasms; Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: stereotacitic body radiation therapy — The patients were treated with high-dose and low fractionated radiotherapy, using modern precision radiotherapy technology.

SUMMARY:
The reirradiation of thoracic tumor is difficult. The possibility of surgery or re course radiotherapy is very small. In the NCCN guideline, only systemic treatment is recommended. However, the effective rate of systemic treatment is low. SBRT has the characteristics of high dose in tumor target area and low dose in surrounding normal tissues. In theory, SBRT is more conducive to the protection of normal tissues and can potentially be used in the salvage treatment of recurrent lesions after radiotherapy. Even so, SBRT is still controversial in the rescue treatment of recurrent lung cancer after radiotherapy, especially for "ultral-central" lesions close to mediastinal structures (such as bronchus, esophagus and large blood vessels), which have a high probability of fatal side effects. However, a few studies on the application of SBRT in the reirradiation for ultral-central lung cancer have shown acceptable safety and efficacy. Generally speaking, there are few studies on SBRT in the treatment of recurrent ultral-central tumor with limited data. The purpose of this study is to further evaluate the efficacy and toxicities of SBRT in the treatment of recurrent ultral-central tumors after radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Pathological diagnosis is malignant tumor.
* The location of the target lesion belongs to the ultra-central type of chest.
* The target lesion had a history of radiotherapy, and the lesion diameter is ≤ 5cm.
* There is no extensive systemic metastasis or although there is metastasis, the metastasis have been controlled by previous treatment.
* KPS>70, no serious or uncontrolled underlying diseases, such as severe or uncontrolled hypertension, diabetes, cardiovascular and cerebrovascular diseases and organ dysfunction, and patients are expected to be tolerated by radiotherapy.

Exclusion Criteria:

* Poor basic pulmonary function or symptom correlation caused by various reasons, unable to lie flat or cooperate with treatment.
* The general condition is poor, and the expected survival time is less than 3 months.
* Psychiatric patients or poor compliance, unable to cooperate to complete treatment.
* For other reasons, the researcher believes that it is not suitable to participate in this trial.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with recurrent chest "ultral-central" malignant tumors after radiotherapy who received SBRT treatment in our department from 2022 to 2023 were expected to be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Toxcicties | From the beginning of the treatment to 3 years after the treatment.
  Adverse events of radiation of normal tissues (Including lung, trachea, bronchus, esophagus, blood vessels, ribs, spinal cord, brachial plexus).
Local control time | From the beginning of the treatment to 3 years after the treatment.
  The time from the date of SBRT to the date of recurrence of the target tumor or the date of last observation.

SECONDARY OUTCOMES:
Overall survival time | From the beginning of the treatment to 3 years after the treatment.
  The time from the date of SBRT to the date of death from any cause or the date of last observation.
Disease progression time | From the beginning of the treatment to 3 years after the treatment.
  The time from the date of SBRT to the date of disease progression from any cause or the date of last observation.

CONTACTS AND LOCATIONS:
Overall Officials: Junjie Wang, M.D., Principal Investigator — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcome measures will be made available.
Supporting Information: CSR
Time Frame: Data will be available within 6 months of the study completion.
Access Criteria: Data access requests will be reviewed by an external Independent Review Panel. Requestors will be required to sign a Data Access Agreement.